CLINICAL TRIAL: NCT07401277
Title: Actinic Keratoses Treated With 5-fluorouracil Plus Aluminum: an Exploratory Study
Brief Title: Actinic Keratoses Treated With 5-fluorouracil Plus Aluminum
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Joanna Kolodney, Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2501092203
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; Powders; Aluminum Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Containers labeled A or B; identity of SOC 5% 5-FU vs investigational 5% 5-FU + 15% ACH concealed from participants and investigators.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Split-Scalp: Left Investigational / Right SOC (Experimental): Participants clinically diagnosed with actinic keratoses (AKs) on the scalp will apply investigational cream (5% 5-fluorouracil [5-FU] + 15% acetyl cysteine [ACH]) to AK lesions on the left half of the scalp and standard of care (SOC) cream (5% 5-FU) to AK lesions on the right half of the scalp. Assignment is determined by sealed, randomized envelopes indicating "Container A to left" (with Container B to right); the identity of A vs B (SOC vs investigational) is blinded to participants and investigators.
  Interventions: Drug: 5% 5-fluorouracil (5-FU) powder; Drug: 5% 5-fluorouracil (5-FU) powder PLUS 15% Aluminum Chloride Hexahydrate (ACH)
- Split-Scalp: Left SOC / Right Investigational (Experimental): Participants clinically diagnosed with AKs on the scalp will apply SOC cream (5% 5-FU) to AK lesions on the left half of the scalp and investigational cream (5% 5-FU + 15% ACH) to AK lesions on the right half of the scalp. Assignment is determined by sealed, randomized envelopes indicating "Container A to right" (with Container B to left); the identity of A vs B (SOC vs investigational) is blinded to participants and investigators.
  Interventions: Drug: 5% 5-fluorouracil (5-FU) powder; Drug: 5% 5-fluorouracil (5-FU) powder PLUS 15% Aluminum Chloride Hexahydrate (ACH)
- Split-Forearm: Left Investigational / Right SOC (Experimental): Participants clinically diagnosed with AKs on the forearms will apply investigational cream (5% 5-FU + 15% ACH) to AK lesions on the left forearm and SOC cream (5% 5-FU) to AK lesions on the right forearm. Assignment is determined by sealed, randomized envelopes indicating "Container A to left" (with Container B to right); the identity of A vs B (SOC vs investigational) is blinded to participants and investigators.
  Interventions: Drug: 5% 5-fluorouracil (5-FU) powder; Drug: 5% 5-fluorouracil (5-FU) powder PLUS 15% Aluminum Chloride Hexahydrate (ACH)
- Split-Forearm: Left SOC / Right Investigational (Experimental): Participants clinically diagnosed with AKs on the forearms will apply SOC cream (5% 5-FU) to AK lesions on the left forearm and investigational cream (5% 5-FU + 15% ACH) to AK lesions on the right forearm. Assignment is determined by sealed, randomized envelopes indicating "Container A to right" (with Container B to left); the identity of A vs B (SOC vs investigational) is blinded to participants and investigators.
  Interventions: Drug: 5% 5-fluorouracil (5-FU) powder; Drug: 5% 5-fluorouracil (5-FU) powder PLUS 15% Aluminum Chloride Hexahydrate (ACH)

INTERVENTIONS:
Drug: 5% 5-fluorouracil (5-FU) powder — Standard of care topical fluorouracil 5% cream, applied twice daily for seven consecutive days to designated side's AK lesions per protocol regimen.
Drug: 5% 5-fluorouracil (5-FU) powder PLUS 15% Aluminum Chloride Hexahydrate (ACH) — Investigational topical combination of fluorouracil 5% and acetyl cysteine 15%, applied twice daily for seven consecutive days to designated side's AK lesions per protocol regimen.

SUMMARY:
Actinic keratoses (AKs) are precancerous skin lesions most common among older white individuals and are prevalent throughout West Virginia. There is a risk of progression to cutaneous squamous cell carcinoma (SCC) when lesions are left untreated. Field-directed therapy with topical agents is used for patients with multiple lesions in a contiguous area. We propose that aluminum utilized for hemostasis is a contributing factor in the tumor regression seen after some biopsies and may be effective as an augmenting agent for topical management of AKs. The primary objective of this study is to determine the effectiveness of using aluminum as an augmenting agent in traditional Standard of Care (SOC) topical cream to treat AKs by assessing the response of AKs to treatment with 5% 5-FU plus 15% aluminum chloride hexahydrate (ACH) cream and comparing the reduction in the number/burden of lesions to SOC topical treatment (5% 5-fluorouracil (5-FU)). Photographs and total counts of AKs will be taken by a single dermatologist before (day 0), immediately after (day 8), and 8 weeks after (day 56) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Less than 50 years due to this being a pathology of adults that develops in chronically sun-damaged skin, individuals <50 years of age are excluded from this study.
* Patients with 4-15 clinically diagnosed AKs on the scalp (16 patients) or on the forearms (16 patients) being followed at the Mohs Surgery clinic by WVU Medicine Dermatology
* Performance status: ECOG Performance status less than or equal to 2
* Patient must provide informed consent

Exclusion Criteria:

* Presence of a suspected squamous cell carcinoma (SCC) or basal cell carcinoma (BCC) lesion or open wound on the treatment site (scalp or forearm)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 15% ACH or other agents used in this study
* Use of one or more of the following products within the past month:

  * Tanning skin colorants
  * Prescription topical drugs
  * Immunomodulatory or immunosuppressive medicines
  * Chemotherapy or cytotoxic medications
  * Photodynamic therapy (PDT) or other treatments of pre-cancers on the skin
  * Vitamin A derivatives taken by mouth
* Patients receiving any other investigational agents
* Patients with immunosuppression or weakened immune systems who may be at a higher risk of infection, including patients who have had chronic lymphocytic leukemia (CLL), who have received transplants, or who are taking medications such as chronic steroids or rheumatoid arthritis (RA) drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Actinic Keratoses; Baseline | Baseline
  Total numerical counts of actinic keratoses (AKs) assessed and documented.
Number of Actinic Keratoses; Day 8 | Day 8
  Total numerical counts of actinic keratoses (AKs) assessed and documented.
Number of Actinic Keratoses; Day 56 | Day 56
  Total numerical counts of actinic keratoses (AKs) assessed and documented.

SECONDARY OUTCOMES:
Skin redness at treatment site(s); Day 8 | Day 8
  Redness will be assessed using a scale of 0-4 as per the Clinical Erythema Assessment grading scale with: 0 = clear, 1 = almost clear, 2 = mild erythema, 3 = moderate erythema, and 4 = severe erythema with 0 being the best outcome.
Skin redness at treatment site(s); Day 56 | Day 56
  Redness will be assessed using a scale of 0-4 as per the Clinical Erythema Assessment grading scale with: 0 = clear, 1 = almost clear, 2 = mild erythema, 3 = moderate erythema, and 4 = severe erythema with 0 being the best outcome.
Skin itchiness at treatment site(s); Day 8 | Day 8
  Itchiness will be assessed using the Peak Pruritus Numeric Rating Scale (NRS) of 0-10 reported by the patient, with 0 being no itchiness and 10 being the worst itchiness ever experienced.
Skin itchiness at treatment site(s); Day 56 | Day 56
  Itchiness will be assessed using the Peak Pruritus Numeric Rating Scale (NRS) of 0-10 reported by the patient, with 0 being no itchiness and 10 being the worst itchiness ever experienced.
Pain at treatment site(s); Day 8 | Day 8
  Pain will be assessed using the Numeric Rating Scale (NRS) of 0-10 reported by the patient, with 0 being no pain and 10 being the worst pain ever experienced.
Pain at treatment site(s); Day 56 | Day 56
  Pain will be assessed using the Numeric Rating Scale (NRS) of 0-10 reported by the patient, with 0 being no pain and 10 being the worst pain ever experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kolodney, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No